CLINICAL TRIAL: NCT01588080
Title: A Pilot Study Comparing Infant Flow SiPAP to Noninvasive NAVA
Brief Title: Comparison Between Infant Flow SiPAP and Noninvasive NAVA in the Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraser Health (Other)
Responsible Party: Principal Investigator, Ravinder Kajla, Respiratory Therapist, Clinical Resource Therapist, Fraser Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAVA
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SiPAP (Placebo Comparator)
  Interventions: Device: SiPAP - placebo
- Neurally Adjusted Ventilatory Assist (Experimental)
  Interventions: Device: Neurally Adjusted Ventilatory Assist (NAVA)

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist (NAVA) — Neurally adjusted ventilatory assist (NAVA), an adjunct that can only be used with the Servo-i ventilator, allows the patient to synchronize spontaneous respiratory effort with mechanical ventilation. NAVA uses the electromyographic signal of the diaphragm (Edi) to transmit this electrical activity back to the ventilator. The NAVA catheter is a functional gastric tube that has electrodes embedded within it and positioned at the level of diaphragm using an electrocardiogram signal. These electrodes continuously (every 5ms) detect the amplitude, duration, and frequency of the Edi and provide pressure support in proportion to this electrical activity. Proportionality is controlled by a NAVA factor (cmH20/microvolt) and is adjusted by the user.
  Arms: Neurally Adjusted Ventilatory Assist
Device: SiPAP - placebo — The Infant Flow® SiPAP provides noninvasive support to neonates. CPAP and Biphasic modes are provided by the Infant Flow® SiPAP. CPAP is an elevated pressure (above atmospheric) and is used to increase a premature babies functional residual capacity (FRC). CPAP is a modality used for babies with both central apneas and mild/moderate increase work of breathing. CPAP increases the FRC and ultimately recruits collapsed alveoli and improves gas exchange in the lungs. BiPhasic, on the other hand, is a modality used for babies that require more respiratory support than CPAP can provide. In BiPhasic mode, respiratory rate (RR), inspiratory time (Ti), and peak inspiratory pressures (PIP) are set and not synchronized with the patients breathing efforts.
  Arms: SiPAP

SUMMARY:
When babies are born premature, they often need help with their breathing. The equipment used to help them breathe is not very comfortable and they sometimes need to be put on a specialized breathing machine with a tube into their lungs. The breathing machine or ventilator can be damaging to the newborn's lungs and more damage can occur the longer the newborn stays on a ventilator leading to chronic lung disease later in their lives. A new device called neurally adjusted ventilatory assist or NAVA is available that the investigators believe may be more comfortable for the premature newborn and may help the baby come off breathing support sooner. When using this device, babies may not need to be put on a ventilator and can avoid the lung damage associated with the breathing tube and the ventilator. The objective of this pilot study is to compare this new breathing device called NAVA, to the equipment that is currently being used, called SiPAP, to support premature newborn's breathing after birth without a breathing tube. The investigators hope to show that with this new technology, premature newborns that are having a difficult time breathing, will come off breathing support sooner compared to the breathing machines that are currently being used. The hypothesis for this proposed study is that improved synchrony with noninvasive NAVA will decrease time spent on noninvasive ventilation and avoid intubation.

ELIGIBILITY:
Inclusion Criteria:

* Infants born greater than or equal to 28+0 weeks and less than or equal to 31+6 weeks gestation
* Diagnosis of RDS in the first 24 hours of life requiring respiratory support
* Parental consent obtained

Exclusion Criteria:

* Infants with a major congenital anomaly
* Infants with pulmonary hypoplasia
* Infants known or suspected to have a neuromuscular disorder
* Infants less than 28+0 weeks GA
* Intubated infants that are likely to require continued mechanical ventilation
* Infants requiring vigorous resuscitation at birth, including chest compressions +/- cardiac medications

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
total duration of respiratory support which includes both days and hours on NAVA/SiPAP (DORS) | one year

SECONDARY OUTCOMES:
Proportion of infants that required escalation to increased noninvasive respiratory support (BiPhasic or increasing NAVA levels) or intubation and mechanical ventilation | one year
All cause mortality during the hospitalization | one year
Bronchopulmonary dysplasia defined as oxygen requirements or ventilatory support needs at 36 weeks CGA | one year
Number of doses of surfactant | one year
Incidence of pneumothorax | one year
Total duration of oxygen requirement | one year
Incidence of nasal deformities, specifically nasal erosions | one year
Time to reach full volume feeds (at least 120 ml/kg/day) | one year
Time to regain birth weight | one year
Total length of hospital stay | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Kajla, Principal Investigator — Fraser Health; Rebecca Sherlock, MD, Study Chair — Fraser Health
Locations (1):
- Surrey Memorial Hospital, Surrey, British Columbia, Canada